CLINICAL TRIAL: NCT03428308
Title: Detection and Treatment of Selected Somatic Chronic Diseases in Patients With Severe Mental Disease: Development and Testing of a Coordinated Interdisciplinary and Intersectoral Intervention
Brief Title: Detection and Treatment of Somatic Disease in Patients With Severe Mental Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Intersectoral Research Unit for Health Services (Other Government)
Collaborators: The City of Copenhagen (Unknown); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Research Unit Of General Practice, Copenhagen (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Anne Marie Lyngsø, Senior researcher, project manager, Intersectoral Research Unit for Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CSU-2017-002
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Ischemia; Cardiac Insufficiency; Diabetes Mellitus, Type 2; Hypertension; Hypercholesterolemia; Severe Mental Disorder
MeSH Terms: conditions — Ischemia; Heart Failure; Diabetes Mellitus, Type 2; Hypertension; Hypercholesterolemia; Mental Disorders | interventions — Mass Screening; Therapeutics

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria will be identified and invited to participate by their general practitioner. Patients who agree to partcipate will be invited to a screening consultation focusing on selected somatic diseases. Patients who are diagnosed with one or more of the selected somatic diseases will be included in the intervention, which consists of individualized courses of treatment focusing on initiation and maintenance of medical treatment and complying with current clinical guidelines and course programmes. The intervention is planned to run for one year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized treatment of detected somatic disease(s) (Experimental)
  Interventions: Other: Screening; Other: Treatment

INTERVENTIONS:
Other: Screening — Each individual general practitioner reviews his/her record system and detects patients who meet the inclusion criteria. Patients who meet these criteria will be invited to participate in the project.
Other: Treatment — Patients who are diagnosed with one or more of the selected somatic diseases receive an individualized course of treatment in general practice, primarily focusing on initiation and maintenance of medical treatment, and complying with current clinical guidelines and course programmes. Treatment goals are set in active co-operation with the patient and his/her family and with supervision and support from the Mental Health Centre Copenhagen, clinical pharmacologists and relevant staff from the municipality in terms of contact/support persons.

SUMMARY:
In Denmark, around 2 % of the population live with severe mental disease. People with severe mental disease live 15-20 years less than the general population. The majority of the years of life lost are a consequence of the excess mortality due to somatic disease. The high prevalence of somatic disease among people with severe mental disease can be largely attributed to physical inactivity, unhealthy diet and side effects from psychopharmacological drugs. Apart from the impacts of unhealthy lifestyle and medication side effects, research suggests that individuals with severe mental disease do not receive the same treatment for their somatic diseases as do the rest of the population. The inequality in diagnostics and treatment can be attributed to stigmatization from healthcare providers and patients' lacking awareness of symptoms and reluctance to seek medical care. Further, the increasing specialization within both somatic and psychiatric care has led to a division between these two treatment systems (8,9). Patients with severe mental disease who simultaneously have one or more somatic diseases need their treatment to be coordinated; such treatment should span general practice, the municipality and the psychiatric and somatic hospital. Accordingly, the following elements are necessary to create effective and coordinated treatment trajectories: detailed preparation, qualitative process evaluation as an integrated part of the courses of treatment, and involvement of all stakeholders from the start.

The overall aim of the project is to optimize the detection of selected chronic somatic diseases, including cardiovascular disease (ischaemia and heart failure), diabetes, hypertension and high cholesterol, in individuals with schizophrenia, schizoaffective disorder or bipolar disorder; to initiate medical treatment; and to ensure treatment compliance among patients.

Accordingly, the project has the following objectives:

* To develop an intervention targeting individuals with schizophrenia, schizoaffective disorder or bipolar disorder that can optimize the detection of selected chronic somatic diseases, including cardiovascular disease (ischaemia and heart failure), diabetes, hypertension and high cholesterol
* To test whether the developed intervention can optimize the detection of cardiovascular disease (ischaemia and heart failure), diabetes, hypertension and high cholesterol in individuals with schizophrenia, schizoaffective disorder or bipolar disorder

The project's hypotheses are that an interdisciplinary and intersectoral intervention targeting individuals with schizophrenia, schizoaffective disorder or bipolar disorder can

* optimize detection of cardiovascular diseases (ischaemia and cardiac insufficiency), diabetes, hypertension and high cholesterol by systematic screening in general practice
* lead to initiation and maintenance of relevant medical treatment. Moreover, we hypothesize that the complete intervention in a long-term perspective will lead to decreased mortality within the target group.

DETAILED DESCRIPTION:
Design, materials and methods:

The project is divided in two phases. In Phase 1 the project's intervention is developed; in Phase 2 the intervention is tested. Phase 2 will be conducted as a feasibility study.

Recruitment:

Based on experience from previous studies, we know the target group can be difficult to recruit and maintain in a course of treatment. We expect that 10-15 patients belonging to each provider-number will meet the project's inclusion criteria. To obtain sufficient patients for the project, we aim to include 20 general practitioners (individual provider-numbers). Accordingly, it is realistic to assume that around 75 patients undergo screening in general practice.

Recruitment of general practitioners will be done by sending written information about project participation and an invitation to participate. Only general practitioners who have one or several practice nurse(s) will be invited. The written invitation will be followed by a telephone call to all invitees to identify those practitioners wishing to participate.

Intervention:

Phase 1: Development of intervention:

The aim of Phase 1 is to design an intervention based on the experiences and perspectives of the involved stakeholders regarding how to optimize detection and treatment of somatic disease among persons with severe mental disease. The project rests on the fundamental idea that it is crucial to involve all relevant stakeholders as early as in the development phase if the intervention is to be effective and feasible to implement in practice. This phase includes 1) meetings with key stakeholders in the field, 2) observations and interviews within the Mental Health Centre Copenhagen and Copenhagen Municipality, 3) multiple project meetings involving all sectors in the project as well as on-going monitoring by the project group.

Phase 2: Testing of the intervention:

The intervention is divided in two parts: a screening intervention and a treatment intervention. The testing of the interventions is conducted as a feasibility study.

Evaluation:

The evaluation is twofold:

1. Evaluation of the effect of the intervention
2. Evaluation of the implementation process

ELIGIBILITY:
Inclusion Criteria:

Patients who appear in their individual general practitioner's record system with one of the following diagnoses:

* Schizophrenia (ICPC code p72)
* Psychosis-schizoaffective disorder without specification (ICPC code p72)
* Bipolar disorder (ICPC code p73)

Exclusion Criteria:

* Persons who live in one of the Municipality of Copenhagen's social-psychiatric residences
* Persons with life-threatening disease
* Persons who do not understand and/or speak the Danish language
* Persons with acute suicidal ideation
* Persons with a severe current abuse incompatible with participation
* Persons who are assessed as being a threat to staff

Ages: 36 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Identified patients with mental disease | Baseline
  Proportion of individuals identified with the selected mental diseases from the general practitioner's total population
Patients attending screening | Baseline
  Proportion of individuals who attend screening out of the total population of individuals who indicate via telephone their wish to participate
Patients diagnosed with somatic disease | Baseline
  Proportion of screened individuals who are diagnosed with one or more of the selected somatic diseases
Patients with untreated somatic disease | Baseline
  Proportion of screened individuals in whom untreated somatic disease is identified
Number of follow-up visits | One year
  Number of follow-up visits for participants in whom medical treatment of somatic disease has been initiated is compared with number of visits in general practice the year before the intervention

SECONDARY OUTCOMES:
Appropriateness of medical treatment | One year
  Whether the patients' medical treatment is appropriate is assessed using the Medication Appropriateness Index (MAI)
Change in HbA1c (blood test) | One year
  Assessment of change in HbA1c since baseline for the participants for whom medical treatment has been initiated
Change in body weight | One year
  Assessment of change in body weight (kilograms) since baseline for the participants for whom medical treatment has been initiated
Change in blood pressure | One year
  Assessment of change in blood pressure (mmHg) since baseline for the participants for whom medical treatment has been initiated
Change in blood cholesterol (blood test) | One year
  Assessment of change in blood cholesterol since baseline for the participants for whom medical treatment has been initiated

OTHER OUTCOMES:
Success of inclusion criteria | One year
  Qualitative interviews with clinicians will be done to assess the success of the inclusion criteria.
Success of exclusion criteria | One year
  Qualitative interviews with clinicians will be done to assess the success of the exclusion criteria.
Success of initiatives for recruiting patients | One year
  Qualitative interviews with clinicians and municipal contact/support persons will be done to assess the success of the process in incentivizing participants to attend screening and subsequent follow-up visits.
  Data registration sheets on attendance and telephonic contact with participants will be evaluated.
Success of screening and treatment | One year
  Qualitative interviews with clinicians and municipal contact/support persons will be done to assess the success of the process in screening and treating the target individuals in general practice
Individual benefits | One year
  Qualitative interviews with clinicians, municipal contact/support persons and participants will be done to assess which individuals benefited from the intervention and which did not.
Circumstances for success | One year
  Qualitative interviews with clinicians, municipal contact/support persons and participants will be done to assess the circumstances under which the intervention succeeded.
Success of intersectoral cooperation | One year
  Qualitative interviews with clinicians, municipal contact/support persons, psychiatrists, clinical pharmacologists and participants will be done to assess how the intersectoral cooperation functioned.

CONTACTS AND LOCATIONS:
Overall Officials: Ane F Bendix, MD, Study Director — Intersectoral Research Unit for Health Services